CLINICAL TRIAL: NCT06776172
Title: Extended Pelvic Lymph Node Dissection vs. No Pelvic Lymph Node Dissection at Radical Prostatectomy in PSMA PET Negative Staged Men: A Multicenter, Randomized Phase III Trial
Brief Title: Extended vs. No Pelvic Lymph Node Dissection During Radical Prostatectomy. DISSECTION 2.0.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02381; bb24Rentsch2; KFS-5775-02-2023 (Other Grant/Funding Number: Krebsforschung Schweiz)
Record Dates: First submitted 2025-01-06; First posted 2025-01-15 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer Surgery; Prostate Cancers
Keywords: Pelvic Lymph Node Dissection
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Radical prostatectomy (RP) with or without pelvic lymph node dissection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical prostatectomy with extended pelvic lymph node dissection (Experimental)
  Interventions: Procedure: Extended Pelvic Lymph Node Dissection
- Radical prostatectomy without extended pelvic lymph node dissection (No Intervention)

INTERVENTIONS:
Procedure: Extended Pelvic Lymph Node Dissection — Extended pelvic lymph node dissection during radical prostatectomy
  Other Names: Extended Lymph Node Dissection
  Arms: Radical prostatectomy with extended pelvic lymph node dissection

SUMMARY:
The aim of the DISSECTION 2.0 study is to determine whether extended pelvic lymph node dissection (ePLND) provides a therapeutic benefit for high-risk prostate cancer patients by improving cancer staging and potentially removing micrometastatic disease, ultimately improving their outcomes.

DETAILED DESCRIPTION:
Prostate cancer is the second most common cancer in men globally and a major cause of cancer deaths in Europe. For men with localized prostate cancer (PCa) and a life expectancy of over 10 years, radical prostatectomy (RP) is the standard treatment. It improves survival compared to conservative management. However, there is debate about de benefit of pelvic lymph node dissection (PLND), the removal of lymph nodes in the pelvis, during RP. While PLND can be omitted in low risk PCa patients, extended PLND (ePLND) is recommended in PCa patients at high-risk for recurrence in order to improve nodal staging The DISSECTION 2.0 study aims to investigate whether extended PLND (ePLND) provides additional benefits for men with high-risk PCa. The hypothesis is that ePLND might help by removing undetectable cancer cells (micrometastases) in the lymph nodes or by better staging the disease for treatment planning. While imaging techniques like PSMA-PET are good at detecting cancer spread, they still miss approximately 60% of cancer-bearing lymph nodes, leaving room for ePLND to potentially improve outcomes.

ePLND involves removing more lymph nodes than standard PLND, leading to better detection of cancer spread. However, it also increases surgery time and complications slightly, though serious complications are rare.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and life expectancy >15 years
* Any biopsy-proven WHO/ISUP grade groups III-V PCa
* High-risk prostate cancer defined as:

  * Any biopsy-proven WHO/ISUP grade group III-V PCa or
  * ISUP grade group II and PSA > 20 ng/ml
* PSMA-PET: negative staging for regional and distant metastasis
* multidisciplinary tumorboard recommendation for radical prostatectomy
* WHO performance status 0-1
* Adequate condition (ASA ≤ III) for general anesthesia and RP

Exclusion Criteria:

* ISUP grade group I PCa and cT1 or cT2 (MRI)
* cT4 (MRI) PCa
* PSMA-PET: positive staging for local and distant metastasis
* Any prior neoadjuvant, local or systemic treatment for PCa
* Previous PLND or pelvic radiotherapy
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence.
* Any other serious underlying medical, psychiatric, psychological, familial, or geographical
* condition, which in the judgment of the investigator may interfere with the planned
* staging, treatment and follow-up, which affect patient compliance or place the patient at
* high risk from treatment-related complications.
* Vulnerable men (participants incapable of judgment or participants under tutelage) will not be included in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2040-02 (Estimated)

PRIMARY OUTCOMES:
Prostate specific antigen (PSA) persistence | 3 month (+/- 2 weeks) postoperatively
  defined as failure to reach a PSA value of <0.1 ng/ml
Biochemical recurrence free survival (BCRFS) | within 24 months post surgery
  time from randomization to biochemical recurrence, defined as serum PSA level ≥ 0.2 ng/ml

SECONDARY OUTCOMES:
PSA persistence (PSAP) above detection limit | postoperative to the end of the study at 10-15 years
  cut-off ≥ 0.03 ng/ml
Initiation time of adjuvant or salvage therapies | postoperative to the end of the study at 10-15 years
  Calculated from randomization to the start of any adjuvant or salvage therapy.
  Salvage radiotherapy (SRT) to the prostatic fossa only excluding lymphatics and without androgen deprivation therapy) will not count as an event for this endpoint if:
  * A PSMA-PET-computed tomography prior to SRT was negative for disease beyond the prostatic fossa, and
  * the SRT led to a PSA <0.1 ng/ml (PSAP) or ≤ 0.2 ng/ml (biochemical recurrence-free survival, BCRFS), respectively.
Time to loco-regional recurrence | from randomization to end of study at 10-15 years
  Calculated from randomization until the first local (prostate bed) or regional (within the extent of the ePLND template) recurrence.
Localization of progression | from randomization to end of study at 10-15 years
  Prostate-specific membrane antigen positron emission tomography (PSMA-PET)
Time to distant metastasis | postoperative to the end of the study at 10-15 years
  Calculated from randomization until the first occurrence of distant metastasis.
Prostate cancer-specific survival | postoperative to the end of the study at 10-15 years
  death due to prostate cancer
Overall survival | postoperative to the end of the study at 10-15 years
  death from any cause
Intraoperative complications | during surgery
  Documented using the CLASSintra classification
Postoperative complications | postoperative up to 10-15 years
  Assessed using the Clavien-Dindo classification
Adverse events (AEs) related to ePLND | postoperative up to 10-15 years
  Categorized according to CTCAE version 5.0
Patient-reported outcome measures (PROMs) | postoperative up to 10-15 years
  tracked using the Expanded Prostate Cancer Index Composite (EPIC)-26 questionnaire Score 1-100 (100 indicates best quality of life score)

OTHER OUTCOMES:
Evaluation of risk prediction for nodal invasion | postoperative to the end of the study at 10-15 years
  from prostate biopsy results
Evaluation of the potential value of unilateral ePLND | postoperative to the end of the study at 10-15 years

CONTACTS AND LOCATIONS:
Locations (15):
- Switzerland (15):
  - Cantonal Hospital Aarau, Aarau
  - University Hospital Basel, Basel
  - Inselspital, Bern
  - Lindenhof Hospital, Bern
  - Cantonal Hospital Biel, Biel
  - Cantonal Hospital Chur, Chur
  - University Hospital Geneva, Geneva
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne
  - Cantonal Hospital Liestal, Liestal
  - Cantonal Hospital Luzern, Lucerne
  - Ospedale Regionale di Lugano, Lugano
  - Cantonal Hospital Neuchâtel, Neuchâtel
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - Hospital Triemli, Zürich, Zurich
  - University Hospital Zürich, Zurich